CLINICAL TRIAL: NCT03512548
Title: A Phase 1, Open-Label, Single-Sequence Crossover Study in Healthy Subjects to Determine the Effect of an Inhibitor of Cytochrome P450 3A on Exposure to Relacorilant and Its Main Metabolites
Brief Title: Study in Healthy Subjects to Determine the Effect of an Inhibitor on Exposure to Relacorilant and Its Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CORT125134-124
Record Dates: First submitted 2018-04-03; First posted 2018-04-30 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — relacorilant; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Period 1 (Experimental): Part 1 Period 1: Relacorilant 350mg will be given once on Day 1
  Interventions: Drug: Relacorilant 350mg
- Part 1 Period 2 (Experimental): Part 1 Period 2: Itraconazole 200mg will be given for three days
  Interventions: Drug: Itraconazole
- Part 1 Period 3 (Experimental): Part 1 Period 3: Relacorilant 350mg will be given once with concomitant itraconazole and itraconazole will continue for three additional days
  Interventions: Drug: Relacorilant 350mg; Drug: Itraconazole
- Part 2 Period A (Experimental): Part 2 Period A: Relacorilant 300mg will be given once daily for 10 days
  Interventions: Drug: Relacorilant 300mg
- Part 2 Period B (Experimental): Part 2 Period B: Relacorilant 300mg will be given once daily in combination with itraconazole 200mg once daily for 10 days
  Interventions: Drug: Itraconazole; Drug: Relacorilant 300mg

INTERVENTIONS:
Drug: Relacorilant 350mg — Relacorilant 350mg
  Other Names: CORT125134
  Arms: Part 1 Period 1; Part 1 Period 3
Drug: Itraconazole — Itraconazole 200 mg
  Other Names: Sporanox
  Arms: Part 1 Period 2; Part 1 Period 3; Part 2 Period B
Drug: Relacorilant 300mg — Relacorilant 300mg
  Other Names: CORT125134
  Arms: Part 2 Period A; Part 2 Period B

SUMMARY:
This is an open label, single sequence, crossover study. In Part 1, eligible subjects will participate in 3 treatment periods, in which they will receive the following treatments in turn: 1) In Period 1, a single 350-mg dose of relacorilant administered alone, 2) In Period 2, once daily 200-mg doses of itraconazole administered for 3 days; 3) In Period 3, single 350-mg dose of relacorilant administered with a concomitant 200-mg dose of itraconazole and continued once daily 200-mg doses of itraconazole for three additional days.

If Part 2 is conducted, eligible subjects will participate in 2 treatment periods, in which they will receive the following treatments in turn: 1) In Period A, once daily 300-mg doses of relacorilant alone for 10 days; 2) In Period B, once daily 300-mg doses of relacorilant in combination with once daily 200-mg doses of itraconazole for 10 days.

DETAILED DESCRIPTION:
This is an open label, single sequence, crossover study. In Part 1, eligible subjects will participate in 3 treatment periods, in which they will receive the following treatments in turn: 1) In Period 1, a single 350-mg dose of relacorilant administered alone, 2) In Period 2, once daily 200-mg doses of itraconazole administered for 3 days; 3) In Period 3, single 350-mg dose of relacorilant administered with a concomitant 200-mg dose of itraconazole and continued once daily 200-mg doses of itraconazole for three additional days.

Part 2 of the study may be conducted if the results of Part 1 indicate that itraconazole has a clinically meaningful effect on exposure to relacorilant and metabolites. If Part 2 is conducted, eligible subjects will participate in 2 treatment periods, in which they will receive the following treatments in turn: 1) In Period A, once daily 300-mg doses of relacorilant alone for 10 days; 2) In Period B, once daily 300-mg doses of relacorilant in combination with once daily 200-mg doses of itraconazole for 10 days.

Blood samples will be collected before dosing and at intervals up to 96 hours after relacorilant dose in Part 1, and up to 24 hours after the last dose of relacorilant in each study period in Part 2. In Part 1 only, additional samples will be collected during the itraconazole dosing to confirm exposure.

Safety and tolerability will be monitored using AEs, clinical laboratory evaluations, 12-lead ECG recordings, vital signs, and and physical examinations.

Subjects will be admitted to the Clinical Research Unit (CRU) on the morning of Day -1 following an 8-hour fast for baseline assessments and will remain confined until completion of procedures. Each subject will have a follow-up (FU) visit 14 ± 2 days (Part 1) or 7 ± 2 days (Part 2) after the last dose of relacorilant.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and risks of the study; willing and able to adhere to scheduled visits, treatment plans, laboratory tests, and other study evaluations and procedures.
2. Give written informed consent.
3. Be males or nonpregnant, nonlactating females judged to be in good health, based on the results of medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory findings.
4. Have a body mass index (BMI) between 18 and 32 kg/m2, inclusive, and a body weight more than 50 kg (110 pounds).
5. Be a nonsmoker. Use of nicotine or nicotine-containing products must be discontinued at least 90 days prior to the first dose of study drug.
6. Be willing to comply with study restrictions
7. Have suitable veins for multiple venipuncture/cannulation.
8. Female subjects must be either of nonchildbearing potential (ie, postmenopausal or permanently sterilized) or use highly effective contraception with low user-dependency.

   * The only acceptable method of highly effective contraception with low user-dependency is an intrauterine device (IUD). Use of hormonal contraception (by any route, including intrauterine hormone releasing systems) or hormone replacement therapy is NOT acceptable.

Exclusion Criteria:

1. Be an employee or immediate family member of the Clinical Research Unit or Corcept.
2. Have been previously enrolled in any study of relacorilant.
3. Have multiple drug allergies, or be allergic to any of the components of Relacorilant and/or itraconazole.
4. Have a condition that could be aggravated by glucocorticoid blockade (eg, asthma, any chronic inflammatory condition).
5. Have a history of malabsorption syndrome or previous gastrointestinal surgery, with the exception of appendectomy and cholecystectomy, which could affect drug absorption or metabolism.
6. Current alcohol or substance abuse.
7. In the 2 calendar months before first study drug administration, have donated/lost blood or plasma in excess of 400 mL.
8. In the 30 days before first study drug administration, have participated in another clinical trial of a new chemical entity or a prescription medicine.
9. Have a positive test for alcohol or drugs of abuse at screening or first admission.
10. Have clinically relevant abnormal findings on vital signs, physical examination, laboratory screening tests, or 12-lead ECG, at screening and/or before first study drug administration, including but not limited to**:

    1. QT interval corrected for heart rate (QTc) using Fridericia's equation (QTcF) >450 ms (from mean of 3 supine ECGs, performed at least 2 minutes apart)
    2. Stage 2 or higher hypertension (supine/semi-recumbent systolic blood pressure [SBP] >160 mmHg, diastolic blood pressure [DBP] >100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart)
    3. Stage 1 hypertension (supine/semi-recumbent SBP 140-160 mmHg, DBP 90-100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart) associated with indication for treatment ie, evidence of end-organ damage, diabetes, or a 10-year cardiovascular risk, estimated using a standard calculator, (eg, QRISK2-2016) greater than 20%
    4. Glomerular filtration rate, estimated using the chronic kidney disease epidemiology (collaboration) (CKD-EPI) method (eGFR; Levey 2009) <60 mL/minute/1.73 m2
    5. Hypokalemia (potassium below lower limit of normal)
    6. Alanine aminotransferase (ALT), aspartate amino transferase (AST), and/or gamma- glutamyltransferase (GGT) >1.5 times the upper limit of normal (ULN)
    7. Seropositive for hepatitis B, hepatitis C, or human immunodeficiency (HIV) viruses **For purposes of qualifying any given subject for study participation, out-of-range values may be repeated once.
11. Have any medical or social reasons for not participating in the study raised by their primary care physician.
12. Have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator.
13. Taken any prohibited prior medication within protocol designated timeframes, such as or including any glucocorticoid, strong inducers, inhibitors or substrates of CYP enzymes involved in drug-drug-interactions, hormonal contraception or hormone replacement therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve up to the last quantifiable sample (AUC0-tz) | predose to 96 hrs postdose in Part 1 and predose to 24 hrs after last dose in Part 2
  Ratio of population geometric means (GMR) for Reference (following oral administration of relacorilant alone) and Test (following the same dose given to subjects concomitantly with itraconazole) areas under plasma concentration-time curve up to the last quantifiable sample (AUC0-tz)

SECONDARY OUTCOMES:
Area under plasma concentration-time curve extrapolated to infinity (AUCinf) | predose to 96 hrs postdose in Part 1; AUCinf not calculated in Part 2 due to steady state evaluation
  Ratio of population geometric means (GMR) for Reference (following oral administration of relacorilant alone) and Test (following the same dose given to subjects concomitantly with itraconazole) areas under plasma concentration-time curve extrapolated to infinity (AUCinf)
Maximum plasma concentration (Cmax) | predose to 96 hrs postdose in Part 1 and predose to 24 hrs after last dose in Part 2
  Ratio of population geometric means (GMR) for Reference (following oral administration of relacorilant alone) and Test (following the same dose given to subjects concomitantly with itraconazole) maximum plasma concentration (Cmax).
Number and Severity of Treatment Emergent Adverse Events | up to 7 weeks in Part 1 and up to 7 weeks in Part 2
  Treatment Emergent Adverse Events will be summarized overall and by treatment based on their frequency and severity of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, PhD, Study Director — Corcept Therapeutics
Locations (1):
- Celerion, Tempe, Arizona, United States